CLINICAL TRIAL: NCT05455138
Title: Allografts in Surgery of the Main Arteries
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ryazan State Medical University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4
Record Dates: First submitted 2022-07-04; First posted 2022-07-13 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Critical Lower Limb Ischemia
Keywords: Critical Lower Limb Ischemia; atherosclerosis; peripheral arterial disease
MeSH Terms: conditions — Atherosclerosis; Peripheral Arterial Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Arterial bypass procedures using autologous venous graft (Experimental): Patients with critical lower limb ischemia due to atherosclerotic peripheral arterial disease who undergo arterial bypass procedures using autologous venous graft
  Interventions: Procedure: Arterial bypass grafting
- Arterial bypass procedures using allogeneic venous graft (Experimental): Patients with critical lower limb ischemia due to atherosclerotic peripheral arterial disease who undergo arterial bypass procedures using allogeneic venous graft
  Interventions: Procedure: Arterial bypass grafting
- Arterial bypass procedures using allogeneic arterial graft (Experimental): Patients with critical lower limb ischemia due to atherosclerotic peripheral arterial disease who undergo arterial bypass procedures using allogeneic arterial graft
  Interventions: Procedure: Arterial bypass grafting
- Arterial bypass procedures using biologic bovine decellularized arterial graft (Experimental): Patients with critical lower limb ischemia due to atherosclerotic peripheral arterial disease who undergo arterial bypass procedures using biologic bovine decellularized arterial graft
  Interventions: Procedure: Arterial bypass grafting

INTERVENTIONS:
Procedure: Arterial bypass grafting — Arterial bypass grafting in patients with critical limb ischemia due to peripheral artery disease

SUMMARY:
The study will examine the results of the use of biological materials (allogeneic arterial grafts, allogeneic venous graft, autologous vein, biological bovine decellularized graft) as a bypass grafts for reconstructive interventions in patients with critical lower limb ischemia due to atherosclerotic peripheral arterial disease in the short-term and long-term postoperative periods. Histological analysis of allogeneic grafts will be carried out at various time points of graft preservation with a Roswell Park Memorial Institute 1640 cell medicum with 400mcg/ml gentamicin and 20mcg/ml fluconazole at a temperature of +4C.

The physical properties of allogeneic grafts from postmortem donors (tensile and tear strength) will be evaluated at various conservation time periods (1 week, 2 weeks, 3 weeks, 4 weeks, 5 weeks, 6 weeks). Markers of endothelial dysfunction (IL-6, endothelin-1, 6-keto-prostaglandin F1alfa, eNOS) will be evaluated in patients with critical ischemia who undergo bypass procedures with arterial and venous allografts at various time points (before surgery, 7 days, 1 month, 3 months, 6 months, 1 year after).

DETAILED DESCRIPTION:
The study will include 200 patients of similar age, gender, and ethnicity, who will be divided into four groups:

Group I: 50 patients who undergo arterial bypass procedures using autologous venous graft derived from great saphenous vein; Group II: 50 patients who undergo arterial bypass procedures using allogeneic venous grafts; Group III: 50 patients who undergo arterial bypass procedures using allogeneic arterial grafts; Group IV: 50 patients using biological bovine decellularized grafts.

Patients will be monitored for 2 years: at inclusion, and 1, 3, 6, 12, 18, and 24 months after bypass procedures.

The primary endpoint of the study will be mortality, i.e. death of the patient from any cause. Secondary endpoints of the study will be graft thrombosis and cardiovascular events such as myocardial infarction, acute coronary syndrome, transient ischemic attack, and stroke.

ELIGIBILITY:
Inclusion Criteria:

* males or females over 18 years of age;
* critical lower limb ischemia due to atherosclerotic peripheral arterial disease.

Exclusion Criteria:

* males or females less than 18 year of age;
* decompensated concomitant pathology;
* pregnancy or lactation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with lethal outcomes | 24 months
  The primary outcome measure is mortality rate

SECONDARY OUTCOMES:
Number of Participants with Graft thrombosis | 24 months
  The secondary outcome measure is graft thrombosis
Myocardial infarction | 1, 3, 6, 12, 18, and 24 months
  The secondary outcome measure is myocardial infarction
Number of Participants with Acute coronary syndrome | 24 months
  The secondary outcome measure is acute coronary syndrome
Number of Participants with Stroke or transient ischemic attack | 24 months
  The secondary outcome measure is stroke or transient ischemic attack

CONTACTS AND LOCATIONS:
Overall Officials: Igor Suchkov, PhD, DMedSc, Principal Investigator — Ryazan State Medical University
Locations (1):
- Ryazan State Medical University, Ryazan, Russia

IPD SHARING:
Plan to Share IPD: No